CLINICAL TRIAL: NCT01287351
Title: Retrospective, Real-life Observational Evaluation of the Effectiveness and Cost-effectiveness of Extra-fine Hydrofluoroalkane (HFA) Beclometasone (BDP) Compared With Fluticasone Propionate (FP) in the Management of Asthma in a Representative Population in the United States (US)
Brief Title: Real-world Effectiveness and Cost-effectiveness of Qvar Versus FP, a US Study
Acronym: USQvarAsthma
Status: Completed | Type: Observational
Sponsor: Research in Real-Life Ltd (Network)
Collaborators: i3 Research (Industry); Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Principal Investigator, David Price, Prof., MD, Professor David Price, Research in Real-Life Ltd
Other Study IDs: 002/10
Record Dates: First submitted 2011-01-28; First posted 2011-02-01 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-08

CONDITIONS: Asthma
Keywords: Real-world; observational; Fluticasone propionate; Metred dose inhaler; Extra-fine hydrofluoroalkane; Asthma management; Inhaled corticosteroids; Beclomethasone dipropionate; USA
MeSH Terms: conditions — Asthma | interventions — Beclomethasone; Fluticasone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- IPDI: Qvar: ICS initiation as Qvar
  Interventions: Drug: extra-fine hydrofluoroalkane beclometasone dipropionate
- IPDI FP: ICS initiation as fluticasone
  Interventions: Drug: Fluticasone propionate
- IPDA Qvar: ICS step-up as Qvar
  Interventions: Drug: extra-fine hydrofluoroalkane beclometasone dipropionate
- IPDA FP: ICS step-up as fluticasone
  Interventions: Drug: Fluticasone propionate

INTERVENTIONS:
Drug: extra-fine hydrofluoroalkane beclometasone dipropionate
  Other Names: Qvar®
  Groups: IPDA Qvar; IPDI: Qvar
Drug: Fluticasone propionate
  Groups: IPDA FP; IPDI FP

SUMMARY:
This study will compare the absolute and relative effectiveness and cost-effectiveness of asthma management in patients in the USA on inhaled corticosteroid (ICS) maintenance therapy as HFA-BDP (Qvar®) pressurised metered dose inhaler (pMDI) compared with fluticasone propionate (FP) pMDI. .

DETAILED DESCRIPTION:
Current asthma guidelines are underpinned by evidence derived from randomised controlled trials (RCTs). Although RCT data are considered the gold standard, patients recruited to asthma RCTs are estimated to represent only a small percentage of the real-world asthma population. The poor representation of the asthma population is due to a number of factors, such as tightly-controlled inclusion criteria for RCTs. There is, therefore, a need to carry out real-world observational studies to inform existing guidelines on the effectiveness of available treatments as used in every-day clinical practice in the heterogeneous asthma population.

Asthma management guidelines recommend long-term, daily anti-inflammatory controller therapy to attenuate the chronic airway inflammation of persistent asthma. The choice of inhaled corticosteroid can be guided by practical considerations (e.g., cost factors) as RCTs have so far failed to identify consistent, significant differences in outcomes among the available inhaled corticosteroids, and data from observational studies are lacking.

FP and HFA-BDP are the two main ICS therapies prescribed in the US for the management of asthma. FP is approximately twice as potent and efficacious, on a microgram basis, as BDP. In clinical trials, however, the extra-fine hydrofluoroalkane (HFA) formulation of BDP has demonstrated potency similar to that of FP. This is felt to be because HFA-BDP shows higher and more even lung deposition than FP, with HFA-BDP, unlike FP, having distribution to both large and small airways.

Owing to similarity of effectiveness of extra-fine HFA-BDP and FP suggested by clinical trial data, and the even lung distribution afforded by the smaller HFA aerosol particles, we hypothesises that extra-fine HFA-BDP may be at least as effective as FP in real-world clinical practice. This hypothesis was supported by a retrospective database study of HFA-BDP versus FP using the UK's General Practice Research Database (GPRD). The study found significantly lower odds for achieving the composite proxy measure for asthma control with FP in both patients initiating ICS therapy (0.77, 95%CI 0.61-0.98) and stepping-up ICS therapy (0.82, 95%CI 0.44-1.52) relative to HFA-BDP. The analysis also revealed that FP was prescribed at significantly higher doses than extra-fine HFA-BDP yet had lower associated odds of achieving asthma control.

In addition to significant health benefits, delivering effective asthma control is critical to reducing the substantial economic burden of asthma, with research indicating annual costs are disproportionately attributable to patients with poorly controlled disease. Recent estimates place the annual figure at 56 billion dollars ($) in the US alone, consisting of direct costs and productivity losses.It is therefore of particular importance to consider outcomes achieved in relation to costs incurred when assessing overall benefit of asthma therapies, with a cost-effectiveness analysis of HFA BDP and FP planned as part of the current study.

The aim of this study is to compare the absolute and relative effectiveness and cost-effectiveness of asthma management in patients in the US on inhaled corticosteroid (ICS) maintenance therapy as extra-fine HFA-BDP (Qvar®) pressurised metered dose inhaler (pMDI) compared with fluticasone propionate (FP) pMDI to further examine the findings of the UK study, and to identify similarities or differences in effectiveness and cost-effectiveness outcomes and prescribing practice between the two countries.

ELIGIBILITY:
Inclusion Criteria:

* Aged: 5-80 years:

  * Paediatric cohort (aged 5-11 years), and
  * Adult cohort (aged 12-60 years)
  * Non-smokers aged 61-80 years
* Evidence of asthma:

  * a diagnostic code for asthma, (ICD 9 codes: 493xx) or
  * ≥2 prescriptions for asthma at different points at any time
* Be on current asthma therapy

  * ≥1 other asthma prescription during the outcome period
* Have at least one year of baseline data (prior to the IPD) and at least one year of outcome data (following the IPD).

Exclusion Criteria:

* had been diagnosed with any chronic respiratory disease at any time other than asthma
* received maintenance oral steroid therapy during baseline.

Updated inclusion criteria - used in the latest analysis:

* Aged 12-60 years (paediatrics included in original study - removed to make comparable with USA data)
* Evidence of asthma: a diagnostic code of asthma or ≥2 scripts for asthma in baseline year at different points in time
* Have definite dosing instructions
* Have at least 1 year of up-to-standard (UTS) baseline data before IPD
* Have at least 1 year of UTS outcome data after IPD. Index dates from 1998 onwards were accepted in the study.

Updated exclusion criteria - used in the latest analysis:

* Had a diagnostic read code for chronic obstructive pulmonary disease (COPD) at any time
* Had a diagnostic read code for chronic respiratory disease at any time
* Were on maintenance oral steroid therapy at baseline

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Asthma patients who either:
  (i) Initiate ICS therapy as one of:
  * HFA-BDP pMDI
  * FP pMDI
  OR
  (ii) Step up ICS therapy as one of:
  * HFA-BDP pMDI
  * FP pMDI
Sampling Method: Non-Probability Sample
Enrollment: 82903 (Actual)
Dates: Start 2004-01; Primary Completion 2008-12 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Proxy Asthma Control | One-year outcome period
  1. No recorded hospital attendance for asthma, including admission, Emergency Room (ER) attendance or Out-Patient Department (OPD) attendance, AND
  2. No prescriptions for acute courses of oral steroids, AND
  3. No GP consultations, hospital admissions or ER attendance for lower respiratory tract infections (LRTI) requiring antibiotics.
Total number of asthma exacerbations and exacerbation rate ratio | One-year outcome period
  Where exacerbations are defined as an occurrence of:
  1. Unscheduled hospital admissions / Emergency Room attendance for asthma, OR
  2. Use of acute courses of oral steroids
Revised proxy asthma control | One-year outcome period
  No recorded hospital attendance for asthma, including admission, Emergency Room (ER) attendance, out-of-hours attendance, or Out-Patient Department (OPD) attendance, AND No prescriptions for acute courses of oral steroids, AND No GP consultations, hospital admissions or ER attendance for lower respiratory tract infections (LRTI) requiring antibiotics.
  Average daily, prescribed dose of ≤180mcg salbutamol / albuterol or ≤500mcg terbutaline
Risk Domain Asthma Control (in the subgroup of patients aged 12-60, the following additional analysis was done) | One year outcome period
  Where control is defined as the absence of the following during the one-year outcome period:
  1. Asthma-related :
     * Hospital attendance or admission, OR
     * A&E attendance, OR
     * Out of hours attendance, OR
     * Out-patient department attendance
  2. GP consultations for lower respiratory tract infection
  3. Prescriptions for acute courses of oral steroids.

SECONDARY OUTCOMES:
Asthma control plus no additional or change in therapy | One-year outcome period
  Success: defined as the absence of
  1. Exacerbation:
     1. Unscheduled hospital admissions / ER attendance for asthma, OR
     2. Acute use of oral steroids
     AND
  2. No consultations, hospital admissions or ER attendance for lower respiratory tract infections (LRTI) requiring antibiotics
     AND
  3. No change in therapeutic regimen:
     1. Increased dose of ICS, and/or
     2. Change in ICS and/or
     3. Change in delivery device, and/or
     4. Use of additional therapy as defined by: long-acting bronchodilator (LABA), theophylline, leukotriene receptor antagonists (LTRAs).
Asthma control plus no additional change in therapy (where change is not driven by possible cost saving) | One-year outcome period
  1. Exacerbation:
     1. Unscheduled hospital admissions / A&E attendance for asthma, OR
     2. Acute use of oral steroids
     AND
  2. No consultations, hospital admissions or A&E attendance for lower respiratory tract infections (LRTI) requiring antibiotics§
     AND
  3. No change in therapeutic regimen:
     1. Increased dose of ICS, and/or
     2. Use of additional therapy as defined by: long-acting bronchodilator (LABA), theophylline, leukotriene receptor antagonists (LTRAs).
Respiratory-related hospitalizations and referrals | One-year outcome period
  Mean number of respiratory-related hospitalizations and referrals per patient during the outcome year
Overall asthma control (Risk and Impairment) (in the subgroup of patients aged 12-60, the following additional analysis was done) | One year outcome period
  Where control is defined as the absence of the following during the one-year outcome period:
  1. Asthma-related :
     * Hospital attendance or admission, OR
     * A&E attendance, OR
     * Out of hours attendance, OR
     * Out-patient department attendance
  2. GP consultations for lower respiratory tract infection
  3. Prescriptions for acute courses of oral steroids.
  AND where the average prescribed daily dose of albuterol or terbutaline is ≤200mg
Health Economic analysis | One year outcome period
  * Drug costs:
    * Short acting beta2 agonist (SABA) costs;
    * Fixed dose combination inhaler costs;
    * Leukotriene receptor antagonists (LTRA) costs;
    * Long acting beta agonists (LABA) costs;
    * Inhaled corticosteroids (ICS) costs;
    * Prednisolone costs;
    * Antibiotics costs;
    * Asthma-related drug costs (including ICS); and
    * Asthma-related drug costs (excluding ICS).
  * Lower respiratory primary care consultation costs;
  * Total respiratory in-patient hospitalisation costs;
  * Total respiratory ER attendance costs;
  * Total respiratory out-patient attendance costs;
  * Other Lower respiratory Medical costs.
Cost-effectiveness analysis | One year outcome period
  Treatment costs will be compared via differences in mean respiratory-related health care costs per patient/year. Treatment effectiveness will be compared via difference in proportion of patients controlled during the outcome period.
  Differences in costs and proportions of patients controlled will be displayed graphically on a cost-effectiveness plane. The four quadrants of the cost-effectiveness plane represent QVAR being:
  * Quadrant I: more costly and more effective (a trade-off);
  * Quadrant II: more costly and less effective (FP dominant);
  * Quadrant III: less costly and less effective (a trade-off); and
  * Quadrant IV: less costly and more effective (QVAR dominant)
  Where the point estimates indicate 'trade-off' between treatments, incremental cost-effectiveness ratio will be calculated:ICER = cQVAR - cFP/eQVAR - eFP (cQVAR and eQVAR are the cost and effectiveness of QVAR respectively and CFP and EFP are the cost and effectiveness of FP).

CONTACTS AND LOCATIONS:
Locations (1):
- Research in Real Life, Cawston, Norfolk, United Kingdom

REFERENCES:
- [Background] Herland K, Akselsen JP, Skjonsberg OH, Bjermer L. How representative are clinical study patients with asthma or COPD for a larger "real life" population of patients with obstructive lung disease? Respir Med. 2005 Jan;99(1):11-9. doi: 10.1016/j.rmed.2004.03.026. PMID 15672843
- [Background] Travers J, Marsh S, Caldwell B, Williams M, Aldington S, Weatherall M, Shirtcliffe P, Beasley R. External validity of randomized controlled trials in COPD. Respir Med. 2007 Jun;101(6):1313-20. doi: 10.1016/j.rmed.2006.10.011. Epub 2006 Nov 17. PMID 17113277
- [Background] Appleton SL, Adams RJ, Wilson DH, Taylor AW, Ruffin RE; North West Adelaide Cohort Health Study Team. Spirometric criteria for asthma: adding further evidence to the debate. J Allergy Clin Immunol. 2005 Nov;116(5):976-82. doi: 10.1016/j.jaci.2005.08.034. PMID 16275363
- [Background] Expert Panel Report 3: Guidelines for the Diagnosis and Management of Asthma. National Heart, Lung, and Blood Institute, National Institutes of Health, 2007. (Accessed March 2008, at http://www.nhlbi.nih.gov/guidelines/asthma/asthgdln.pdf.)
- [Background] British Guideline on the Management of Asthma, May 2008. 2008. (Accessed 26 June 2008, at http://www.sign.ac.uk/guidelines/fulltext/101/index.html.)
- [Background] Global Strategy for Asthma Management and Prevention, updated 2008. 2008. (Accessed at http://www.ginasthma.org.)
- [Background] Fanta CH. Asthma. N Engl J Med. 2009 Mar 5;360(10):1002-14. doi: 10.1056/NEJMra0804579. No abstract available. PMID 19264689
- [Background] Shepherd J, Rogers G, Anderson R, Main C, Thompson-Coon J, Hartwell D, Liu Z, Loveman E, Green C, Pitt M, Stein K, Harris P, Frampton GK, Smith M, Takeda A, Price A, Welch K, Somerville M. Systematic review and economic analysis of the comparative effectiveness of different inhaled corticosteroids and their usage with long-acting beta2 agonists for the treatment of chronic asthma in adults and children aged 12 years and over. Health Technol Assess. 2008 May;12(19):iii-iv, 1-360. doi: 10.3310/hta12190. PMID 18485271
- [Background] Aubier M, Wettenger R, Gans SJ. Efficacy of HFA-beclomethasone dipropionate extra-fine aerosol (800 microg day(-1)) versus HFA-fluticasone propionate (1000 microg day(-1)) in patients with asthma. Respir Med. 2001 Mar;95(3):212-20. doi: 10.1053/rmed.2000.1025. PMID 11266239
- [Background] Fairfax A, Hall I, Spelman R. A randomized, double-blind comparison of beclomethasone dipropionate extrafine aerosol and fluticasone propionate. Ann Allergy Asthma Immunol. 2001 May;86(5):575-82. doi: 10.1016/S1081-1206(10)62907-9. PMID 11379810
- [Background] Lasserson TJ, Cates CK, Jones AB, Steele EH, White J. Fluticasone versus HFA-beclomethasone dipropionate for chronic asthma in adults and children. Cochrane Database Syst Rev. 2006 Apr 19;2006(2):CD005309. doi: 10.1002/14651858.CD005309.pub3. PMID 16625634
- [Background] Teva Pharmaceutical Industries, 2010. Data on file.
- See also: Optimum Patient Care is the Research in Real Life's sister company (a social enterprise organisation) — http://www.optimumpatientcare.org